CLINICAL TRIAL: NCT03975478
Title: BASALTO (Bariatric Surgery and LDL Cholesterol) Trial
Brief Title: Bariatric Surgery and LDL Cholesterol
Acronym: BASALTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/8471/I
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; gastric bypass; sleeve gastrectomy; LDL cholesterol; morbid obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for statistical analysis will be blinded to group allocation until data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric bypass (Active Comparator): Bariatric surgery by gastric bypass (GB)
  Interventions: Procedure: Gastric bypass
- Sleeve gastrectomy (Experimental): Bariatric surgery by sleeve gastrectomy (SG)
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Gastric bypass — The GB technique consists of a 150-cm antecolic Roux limb with a 25-mm circular pouch-jejunostomy and exclusion of 50 cm of the proximal jejunum.
  Arms: Gastric bypass
Procedure: Sleeve gastrectomy — The SG technique consists of a longitudinal resection of the stomach from the angle of His to approximately 5 cm proximal to the pylorus, using a 35 French bougie inserted along the lesser curvature.
  Arms: Sleeve gastrectomy

SUMMARY:
Background:

Observational studies have shown that gastric bypass is superior to sleeve gastrectomy in terms of LDL cholesterol improvement. If these results are confirmed in randomized controlled trials, pre-surgical LDL cholesterol status should be a point to consider in the surgical procedure election.

Objective:

The primary objective is to compare 1-year LDL cholesterol remission after gastric bypass and sleeve gastrectomy in morbid obese patients.

Methods:

Phase 3, uni-centric, randomized clinical trial, with intention-to-treat analysis to compare LDL cholesterol remission between gastric bypass and sleeve gastrectomy with a 12 months follow-up. The inclusion criteria will be patients aged between 18-60 years old with a body mass index ≥40 or ≥35 kg/m2 with a significant obesity related comorbidity and high LDL cholesterol levels. Patients will be evaluated preoperatively (2 months before surgery) and at 3, 6 and 12 months after bariatric surgery. Examinations will include routine blood chemistry, anthropometric measures, food intake recall, physical activity questionnaires,intima media thickness, fecal samples for microbiota examinations, fat tissue samples and serum samples for lipidomics and hormonal analyses.

DETAILED DESCRIPTION:
In the preoperative period, patients will follow a standard nutritional intervention that includes 6 monthly group sessions focused on achieving changes in dietary habits and hence ease adaptation after surgery.

In addition, lipid-lowering treatment will be adjusted and standardized following the Institut Català de la Salut clinical practice guidelines. Cholesterol-lowering drugs will be withdrawn immediately after the surgical intervention to asses LDL cholesterol remission during follow-up.

After surgery, a standardized protocol will be followed for the two groups in relation to dietary recommendations and physical activity, as well as the initiation of lipid-lowering medication after the intervention, in order to avoid the bias that may arise due to an open study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥40 or BMI ≥35 kg/m2 with a significant obesity related comorbidities.
* Age 18 - 60 years.
* Previous successfully instituted and supervised but failed adequate diet and exercise program.
* Elevated LDL cholesterol defined as LDL cholesterol concentration >130 mg/dL or treatment with cholesterol-lowering drugs.

Exclusion Criteria:

* BMI >60 kg/m2.
* Previous BS.
* Exclusion criteria for BS:

  * Significant psychiatric disorder.
  * Severe eating disorder, active alcohol or substance abuse.
  * Contraindications for major abdominal surgery.
  * Active gastric ulcer disease.
  * Severe hepatic diseases.
  * Pregnancy or breastfeeding.
* Cases in whom SG or GB are preferred:

  * Severe symptomatic gastro esophageal reflux disease despite medication.
  * Large hiatal hernia.
  * Expected dense adhesions at the level of the small bowel.
  * Need for endoscopic follow-up of the duodenum, history of inflammatory bowel disease.
  * History of renal transplantation in which drug malabsorption can be caused with a GB.
* Cholesterol lowering drugs will be withdrawn immediately after the surgical intervention to asses LDL cholesterol remission during follow-up. Cases in whom perioperative statins withdrawn cannot be adequate will be excluded:

  * Established cardiovascular disease or subclinical cardiovascular disease (atheroma plaque detection in carotid ultrasonography exam) in which LDL cholesterol objectives are more aggressive or statins can be prescribed independently of LDL cholesterol levels.
  * LDL cholesterol >190 mg/dL or history of familial hypercholesterolemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
LDL cholesterol remission 1 year after GB and SG | At 12 months after surgery
  Postoperative LDL cholesterol <130 mg/dL without cholesterol-lowering drugs

SECONDARY OUTCOMES:
LDL cholesterol remission at 3 months after GB and SG | At 3 months after surgery
  Postoperative LDL cholesterol <130 mg/dL without cholesterol-lowering drugs
LDL cholesterol remission at 6 months after GB and SG | At 6 months after surgery
  Postoperative LDL cholesterol <130 mg/dL without cholesterol-lowering drugs
LDL cholesterol improvement postoperatively | At 12 months after surgery
  In patients without preoperative cholesterol lowering drugs: Decrease ≥20% in LDL cholesterol concentration (mg/dL) without cholesterol-lowering drugs.
  In patients with preoperative cholesterol lowering drugs: Medication withdrawn and LDL cholesterol >130 mg/dL, or decrease ≥20% in LDL cholesterol concentration without medication withdrawn.
Hypertriglyceridemia remission postoperatively | 12 months after surgery
  Triglyceride concentration <150 mg/dL without fibrates
Low HDL cholesterol remission postoperatively | 12 months after surgery
  HDL cholesterol concentration >50 mg/dL in women, or >40 mg/dL in men
Changes in LDL cholesterol concentration postoperatively | At 3 months after surgery
  Variation of LDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in LDL cholesterol concentration postoperatively | At 6 months after surgery
  Variation of LDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in LDL cholesterol concentration postoperatively | At 12 months after surgery
  Variation of LDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in total cholesterol during follow-up | At 3 months after surgery
  Variation of total cholesterol concentration (mg/dL) with respect to preoperative value
Changes in total cholesterol during follow-up | At 6 months after surgery
  Variation of total cholesterol concentration (mg/dL) with respect to preoperative value
Changes in total cholesterol during follow-up | At 12 months after surgery
  Variation of total cholesterol concentration (mg/dL) with respect to preoperative value
Changes in HDL cholesterol during follow-up | At 3 months after surgery
  Variation of HDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in HDL cholesterol during follow-up | At 6 months after surgery
  Variation of HDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in HDL cholesterol during follow-up | At 12 months after surgery
  Variation of HDL cholesterol concentration (mg/dL) with respect to preoperative value
Changes in triglycerides during follow-up | At 3 months after surgery
  Variation of triglycerides concentration (mg/dL) with respect to preoperative value
Changes in triglycerides during follow-up | At 6 months after surgery
  Variation of triglycerides concentration (mg/dL) with respect to preoperative value
Changes in triglycerides during follow-up | At 12 months after surgery
  Variation of triglycerides concentration (mg/dL) with respect to preoperative value
Changes in lipoprotein(a) during follow-up | At 3 months after surgery
  Variation of lipoprotein(a) concentration (mg/dL) with respect to preoperative value
Changes in lipoprotein(a) during follow-up | At 6 months after surgery
  Variation of lipoprotein(a) concentration (mg/dL) with respect to preoperative value
Changes in lipoprotein(a) during follow-up | At 12 months after surgery
  Variation of lipoprotein(a) concentration (mg/dL) with respect to preoperative value
Changes in lipoproteins particle size | At 3 months postoperatively
  Variation of LDL cholesterol particle size (nm) with respect to preoperative value
Changes in lipoproteins composition | At 3 months postoperatively
  Variation of LDL cholesterol particles concentration (nmol/L) with respect to preoperative value
Changes in lipoproteins particle size | At 6 months postoperatively
  Variation of LDL cholesterol particle size (nm) with respect to preoperative value
Changes in lipoproteins composition | At 6 months postoperatively
  Variation of LDL cholesterol particles concentration (nmol/L) with respect to preoperative value
Changes in lipoproteins particle size | At 12 months postoperatively
  Variation of LDL cholesterol particle size (nm) with respect to preoperative value
Changes in lipoproteins composition | At 12 months postoperatively
  Variation of LDL cholesterol particles concentration (nmol/L) with respect to preoperative value
Change in patients' estimated cardiovascular risk | At 3 months postoperatively
  Variation of REGICOR score (10-year estimated cardiovascular risk, %) with respect to preoperative value
Change in patients' estimated cardiovascular risk | At 6 months postoperatively
  Variation of REGICOR score (10-year estimated cardiovascular risk, %) with respect to preoperative value
Change in patients' estimated cardiovascular risk | At 12 months postoperatively
  Variation of REGICOR score (10-year estimated cardiovascular risk, %) with respect to preoperative value
Type 2 diabetes complete remission | At 3 months postoperatively
  Glycated hemoglobin [HbA1c] value <6.0% and fasting glucose level <100 mg/dL without diabetes medications
Type 2 diabetes complete remission | At 6 months postoperatively
  Glycated hemoglobin [HbA1c] value <6.0% and fasting glucose level <100 mg/dL without diabetes medications
Type 2 diabetes complete remission | At 12 months postoperatively
  Glycated hemoglobin [HbA1c] value <6.0% and fasting glucose level <100 mg/dL without diabetes medications
Type of mechanisms involved in the different LDL cholesterol remission rates after GB and SG | At 3 months postoperatively
  Different eligible types: Weight loss, changes in targeted lipidomics, changes in lipoproteins particles size and composition, changes in dietary habits and physical activity, modifications in gut microbiota, gene and protein expression in adipose tissue, changes in gut hormones
Type of mechanisms involved in the different LDL cholesterol remission rates after GB and SG | At 6 months postoperatively
  Different eligible types: Weight loss, changes in targeted lipidomics, changes in lipoproteins particles size and composition, changes in dietary habits and physical activity, modifications in gut microbiota, gene and protein expression in adipose tissue, changes in gut hormones
Type of mechanisms involved in the different LDL cholesterol remission rates after GB and SG | At 12 months postoperatively
  Different eligible types: Weight loss, changes in targeted lipidomics, changes in lipoproteins particles size and composition, changes in dietary habits and physical activity, modifications in gut microbiota, gene and protein expression in adipose tissue, changes in gut hormones
Changes in intima media thickness | At 12 months postoperatively
  Variation of mean intima-media thickness (IMT, in mm) measured ultrasonographically in the far wall of bilateral common carotid arteries with respect to preoperative value

CONTACTS AND LOCATIONS:
Overall Officials: David Benaiges Boix, Dr, Principal Investigator — Hospital del Mar (Barcelona, Spain)
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Allison DB, Fontaine KR, Manson JE, Stevens J, VanItallie TB. Annual deaths attributable to obesity in the United States. JAMA. 1999 Oct 27;282(16):1530-8. doi: 10.1001/jama.282.16.1530. PMID 10546692
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Grundy SM. Obesity, metabolic syndrome, and cardiovascular disease. J Clin Endocrinol Metab. 2004 Jun;89(6):2595-600. doi: 10.1210/jc.2004-0372. No abstract available. PMID 15181029
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Salminen P, Helmio M, Ovaska J, Juuti A, Leivonen M, Peromaa-Haavisto P, Hurme S, Soinio M, Nuutila P, Victorzon M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss at 5 Years Among Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):241-254. doi: 10.1001/jama.2017.20313. PMID 29340676
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Peterli R, Wolnerhanssen BK, Peters T, Vetter D, Kroll D, Borbely Y, Schultes B, Beglinger C, Drewe J, Schiesser M, Nett P, Bueter M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity: The SM-BOSS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):255-265. doi: 10.1001/jama.2017.20897. PMID 29340679
- [Background] Angrisani L, Santonicola A, Iovino P, Vitiello A, Zundel N, Buchwald H, Scopinaro N. Bariatric Surgery and Endoluminal Procedures: IFSO Worldwide Survey 2014. Obes Surg. 2017 Sep;27(9):2279-2289. doi: 10.1007/s11695-017-2666-x. PMID 28405878
- [Background] Arterburn D, Gupta A. Comparing the Outcomes of Sleeve Gastrectomy and Roux-en-Y Gastric Bypass for Severe Obesity. JAMA. 2018 Jan 16;319(3):235-237. doi: 10.1001/jama.2017.20449. No abstract available. PMID 29340659
- [Background] Climent E, Benaiges D, Pedro-Botet J, Goday A, Sola I, Ramon JM, Flores-LE Roux JA, Checa MA. Laparoscopic Roux-en-Y gastric bypass vs. laparoscopic sleeve gastrectomy for morbid obesity: a systematic review and meta-analysis of lipid effects at one year postsurgery. Minerva Endocrinol. 2018 Mar;43(1):87-100. doi: 10.23736/S0391-1977.17.02627-X. Epub 2017 Feb 15. PMID 28206728
- [Background] Casajoana A, Pujol J, Garcia A, Elvira J, Virgili N, de Oca FJ, Duran X, Fernandez-Veledo S, Vendrell J, Vilarrasa N. Predictive Value of Gut Peptides in T2D Remission: Randomized Controlled Trial Comparing Metabolic Gastric Bypass, Sleeve Gastrectomy and Greater Curvature Plication. Obes Surg. 2017 Sep;27(9):2235-2245. doi: 10.1007/s11695-017-2669-7. PMID 28451931
- [Background] Schiavon CA, Bersch-Ferreira AC, Santucci EV, Oliveira JD, Torreglosa CR, Bueno PT, Frayha JC, Santos RN, Damiani LP, Noujaim PM, Halpern H, Monteiro FLJ, Cohen RV, Uchoa CH, de Souza MG, Amodeo C, Bortolotto L, Ikeoka D, Drager LF, Cavalcanti AB, Berwanger O. Effects of Bariatric Surgery in Obese Patients With Hypertension: The GATEWAY Randomized Trial (Gastric Bypass to Treat Obese Patients With Steady Hypertension). Circulation. 2018 Mar 13;137(11):1132-1142. doi: 10.1161/CIRCULATIONAHA.117.032130. Epub 2017 Nov 13. PMID 29133606
- [Background] Pihlajamaki J, Gronlund S, Simonen M, Kakela P, Moilanen L, Paakkonen M, Pirinen E, Kolehmainen M, Karja V, Kainulainen S, Uusitupa M, Alhava E, Miettinen TA, Gylling H. Cholesterol absorption decreases after Roux-en-Y gastric bypass but not after gastric banding. Metabolism. 2010 Jun;59(6):866-72. doi: 10.1016/j.metabol.2009.10.004. Epub 2009 Dec 16. PMID 20015521
- [Background] Hanusch-Enserer U, Zorn G, Wojta J, Kopp CW, Prager R, Koenig W, Schillinger M, Roden M, Huber K. Non-conventional markers of atherosclerosis before and after gastric banding surgery. Eur Heart J. 2009 Jun;30(12):1516-24. doi: 10.1093/eurheartj/ehp108. Epub 2009 Apr 20. PMID 19380349
- [Background] Asztalos BF, Swarbrick MM, Schaefer EJ, Dallal GE, Horvath KV, Ai M, Stanhope KL, Austrheim-Smith I, Wolfe BM, Ali M, Havel PJ. Effects of weight loss, induced by gastric bypass surgery, on HDL remodeling in obese women. J Lipid Res. 2010 Aug;51(8):2405-12. doi: 10.1194/jlr.P900015. PMID 20631298
- [Background] Knopp RH, Gitter H, Truitt T, Bays H, Manion CV, Lipka LJ, LeBeaut AP, Suresh R, Yang B, Veltri EP; Ezetimibe Study Group. Effects of ezetimibe, a new cholesterol absorption inhibitor, on plasma lipids in patients with primary hypercholesterolemia. Eur Heart J. 2003 Apr;24(8):729-41. doi: 10.1016/s0195-668x(02)00807-2. PMID 12713767
- [Background] Samczuk P, Ciborowski M, Kretowski A. Application of Metabolomics to Study Effects of Bariatric Surgery. J Diabetes Res. 2018 Mar 11;2018:6270875. doi: 10.1155/2018/6270875. eCollection 2018. PMID 29713650
- [Background] Ramos-Molina B, Castellano-Castillo D, Alcaide-Torres J, Pastor O, de Luna Diaz R, Salas-Salvado J, Lopez-Moreno J, Fernandez-Garcia JC, Macias-Gonzalez M, Cardona F, Tinahones FJ. Differential effects of restrictive and malabsorptive bariatric surgery procedures on the serum lipidome in obese subjects. J Clin Lipidol. 2018 Nov-Dec;12(6):1502-1512. doi: 10.1016/j.jacl.2018.07.006. Epub 2018 Jul 25. PMID 30143432
- [Background] Buchwald H, Rudser KD, Williams SE, Michalek VN, Vagasky J, Connett JE. Overall mortality, incremental life expectancy, and cause of death at 25 years in the program on the surgical control of the hyperlipidemias. Ann Surg. 2010 Jun;251(6):1034-40. doi: 10.1097/SLA.0b013e3181deb4d0. PMID 20485136
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):e285-e350. doi: 10.1016/j.jacc.2018.11.003. Epub 2018 Nov 10. No abstract available. PMID 30423393
- [Background] Rubino F, Kaplan LM, Schauer PR, Cummings DE; Diabetes Surgery Summit Delegates. The Diabetes Surgery Summit consensus conference: recommendations for the evaluation and use of gastrointestinal surgery to treat type 2 diabetes mellitus. Ann Surg. 2010 Mar;251(3):399-405. doi: 10.1097/SLA.0b013e3181be34e7. PMID 19934752
- [Background] Ciurana Misol R, Franzi Sisó A, García Cerdán MR, Ríos Rodríguez MA, Ramos Blanes R, Solanas Saura P, et al. Guies de pràctica clínica. Colesterol i risc coronari. General Catalunya Inst Català de la Salut. 2009;1-131. Available from: http://www.gencat.cat/ics/professionals/guies/docs/material_docent_colesterol.pdf
- [Background] Buse JB, Caprio S, Cefalu WT, Ceriello A, Del Prato S, Inzucchi SE, McLaughlin S, Phillips GL 2nd, Robertson RP, Rubino F, Kahn R, Kirkman MS. How do we define cure of diabetes? Diabetes Care. 2009 Nov;32(11):2133-5. doi: 10.2337/dc09-9036. No abstract available. PMID 19875608
- [Background] Marrugat J, D'Agostino R, Sullivan L, Elosua R, Wilson P, Ordovas J, Solanas P, Cordon F, Ramos R, Sala J, Masia R, Kannel WB. An adaptation of the Framingham coronary heart disease risk function to European Mediterranean areas. J Epidemiol Community Health. 2003 Aug;57(8):634-8. doi: 10.1136/jech.57.8.634. PMID 12883073
- [Background] Hutter MM, Schirmer BD, Jones DB, Ko CY, Cohen ME, Merkow RP, Nguyen NT. First report from the American College of Surgeons Bariatric Surgery Center Network: laparoscopic sleeve gastrectomy has morbidity and effectiveness positioned between the band and the bypass. Ann Surg. 2011 Sep;254(3):410-20; discussion 420-2. doi: 10.1097/SLA.0b013e31822c9dac. PMID 21865942
- [Background] Climent E, Benaiges D, Flores-Le Roux JA, Ramon JM, Pedro-Botet J, Goday A. Changes in the lipid profile 5 years after bariatric surgery: laparoscopic Roux-en-Y gastric bypass versus laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2018 Aug;14(8):1099-1105. doi: 10.1016/j.soard.2018.05.006. Epub 2018 May 19. PMID 29941302
- [Background] Benaiges D, Goday A, Ramon JM, Hernandez E, Pera M, Cano JF; Obemar Group. Laparoscopic sleeve gastrectomy and laparoscopic gastric bypass are equally effective for reduction of cardiovascular risk in severely obese patients at one year of follow-up. Surg Obes Relat Dis. 2011 Sep-Oct;7(5):575-80. doi: 10.1016/j.soard.2011.03.002. Epub 2011 Mar 17. PMID 21546321
- [Derived] Benaiges D, Lazaro I, Goday A, Sala-Vila A, Haro N, Flores-Le Roux JA, Fito M, Casajoana A, Climent E, Alechaga E, Nebot P, Castaner O, Pedro-Botet J, Pozo OJ. Targeted lipidomics reveals distinct mechanisms driving LDL cholesterol response to gastric bypass and sleeve gastrectomy: An exploratory study. Nutr Metab Cardiovasc Dis. 2026 Jan 13:104567. doi: 10.1016/j.numecd.2026.104567. Online ahead of print. PMID 41622097
- [Derived] Benaiges D, Goday A, Casajoana A, Flores-Le Roux JA, Fito M, Pozo OJ, Serra C, Pera M, Llaurado G, Climent E, Villatoro M, Lazaro I, Castaner O, Pedro-Botet J. Short-term effects of gastric bypass versus sleeve gastrectomy on high LDL cholesterol: The BASALTO randomized clinical trial. Cardiovasc Diabetol. 2024 Jun 15;23(1):205. doi: 10.1186/s12933-024-02296-x. PMID 38879559
- [Derived] Benaiges D, Goday A, Flores-Le Roux JA, Fito M, Pozo O, Rodriguez-Morato J, Serra C, Pera M, Llaurado G, Climent E, Castaner O, Ramon JM, Pedro-Botet J. Bariatric surgery and LDL cholesterol (BASALTO) trial study protocol: randomised controlled study evaluating the effect of gastric bypass versus sleeve gastrectomy on high LDL cholesterol. BMJ Open. 2020 Sep 10;10(9):e037712. doi: 10.1136/bmjopen-2020-037712. PMID 32912989